CLINICAL TRIAL: NCT02039804
Title: Sodium Hyaluronate Injection and Corticosteroids in Trochanteric Bursitis: a Randomized Controlled Study.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Sascha Colen, MD, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Trochanter Bursitis
Record Dates: First submitted 2013-07-24; First posted 2014-01-20 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Adrenal Cortex Hormones; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronic acid (Experimental): Injectable hyaluronic acid.
  Interventions: Device: Hyaluronic acid
- Corticosteroids (Active Comparator): Injectable corticosteroids.
  Interventions: Drug: Corticosteroids

INTERVENTIONS:
Drug: Corticosteroids — Intra-bursal injection
  Other Names: Depo-Medrol 40mg
  Arms: Corticosteroids
Device: Hyaluronic acid — Intra-bursal injection
  Other Names: SportVis
  Arms: Hyaluronic acid

SUMMARY:
Trochanteric pain can be caused by osteoarthritis of the hip, fracture, tendinitis, nerve pathology and trochanteric bursitis. Trochanteric bursitis is often seen at the outpatient clinic and is characterized by chronic lateral hip pain in the vicinity of the trochanter major, overlying the lateral aspect of the hip. When pain is persistent after conventional therapies, anesthetic and corticosteroid (CS) injections can provide short term to intermediate relief of pain, but relapse is common. Only one retrospective study showed the efficacy of intra-bursal trochanteric injections with HA and CS. They concluded that the pain release is significant with large effect sizes for both treatment. However, the efficacy of CS appeared to be short lived and it was shown that the efficacy of HA at 6 and 12 months is significant compared to CS (p<0.05).

In this study we want to compare the efficacy of corticosteroids and hyaluronic acid in the treatment of trochanteric bursitis.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years and older, but <75 years;
* VAS for pain > 30mm;
* Diagnosis of trochanteric bursitis as suggested by Brinks et al with symptoms for more than 3 months (3);
* Failure of conservative therapy of more than one month;
* Written informed consent;
* Available for the duration of the investigation.

Exclusion Criteria:

* Previous surgery in the same region;
* Current other problem(s) in the affected extremity;
* Diabetes mellitus;
* Patient who received a local (CS) injection within 3 months from the baseline visit;
* Allergic or hypersensitive to CS or HA;
* Patients suffering (chronic) low back pain with or without sciatic pain;
* Patients with radiographic signs of moderate or severe hip osteoarthritis (Kellgren and Lawrence >1);
* Pregnant or lactating, or woman of childbearing potential not willing to use an acceptable method of contraception during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
VAS for pain | 26 weeks after administration

SECONDARY OUTCOMES:
Harris Hip Score | 6, 12, 26 weeks
VAS for pain | 6 and 12 weeks after administration

OTHER OUTCOMES:
Patient's Global Assessment of Normal Function/Activity | 6, 12, 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Colen, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium